CLINICAL TRIAL: NCT04701359
Title: Comparison of Cobalt-Chromium (CoCr) Alloy and Titanium-Nitride (TiN) Coating in Total Knee Arthroplasty: A Prospective, Randomised, Double-blinded Clinical Trial
Brief Title: Comparison of CoCr Alloy and TiN Coating in TKA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Implant to be analysed not used at study centre any more.
Sponsor: Medical University of Graz (Other)
Collaborators: Alphamed Medizintechnik Fischer GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1533/2020
Record Dates: First submitted 2020-10-30; First posted 2021-01-08 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Knee; Arthroplasty, Replacement, Knee
Keywords: Implant coating/alloy; Titanium-Nitride (TiN) coating; Cobalt-Chromium (CoCr) alloy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Two-hundred patients with knee osteoarthritis included altogether. Patients randomly assigned to group A (receiving total knee arthroplasty [TKA] with TiN-coating) or group B (receiving TKA with CoCr-alloy).
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking of both patients and outcome assessors. Only care provider (i.e. surgeon) and investigator aware of implant-type used. During follow-up, neither care provider nor investigator allowed to assess patients' study-specific outcome. As implants look identical on X-rays, allocation to one or another group cannot be verified by independent outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (TiN-coating) (Experimental): Patients with knee osteoarthritis receive total knee arthroplasty with Titanium-Nitride (TiN)-coated implant.
  Interventions: Device: TiN-alloy based total knee arthroplasty
- Group B (CoCr-alloy) (Active Comparator): Patients with knee osteoarthritis receive total knee arthroplasty with Cobalt-Chromium (CoCr)-alloy implant.
  Interventions: Device: CoCr-coating based total knee arthroplasty

INTERVENTIONS:
Device: TiN-alloy based total knee arthroplasty — TiN-alloy based TKA implanted for knee osteoarthritis.
  Other Names: ACS System, Implantcast GmbH, Buxtehude, Germany
  Arms: Group A (TiN-coating)
Device: CoCr-coating based total knee arthroplasty — CoCr-coating based TKA implanted for knee osteoarthritis.
  Other Names: ACS System, Implantcast GmbH, Buxtehude, Germany
  Arms: Group B (CoCr-alloy)

SUMMARY:
In the current prospective, randomized study, two different materials of the same total knee arthroplasty (TKA) system - cobalt-chromium (CoCr) and titanium-nitride (TiN) - are going to be compared with regards to postoperative outcome. Two-hundred patients are planned to be included in the study over a 4-year period, randomly assigned to either the CoCr- or TiN-implant-group. In order to ensure double-blinding, patients will not be informed about the group they had been assigned to. Moreover, no identifying information of the implant used will be written on documents later accessible to nurses and/or physicians at follow-up appointments. Consequently, surgeons of the respective patients will be excluded from study-specific examination of patients. Despite range of motion (ROM), questionnaires (visual analogue scale - VAS; Western Ontario and McMaster Universities Osteoarthritis Index - WOMAC, Forgotten Joint Score - FJS; Knee Society Scoe - KSS) will be used to assess the postoperative outcome. Furthermore, metal ion levels (cobalt, chrom, molybdenum, titanium) in the blood stream of patients will be measured at scheduled follow-up appointments. It is expected that there will not be a measureable difference between the two coating-groups with regards to ROM, functionality, and metal-ion levels over time.

DETAILED DESCRIPTION:
Rationale

The present double-blinded study was planned in order to assess whether differences in materials - using one otherwise similar TKA system - would have an effect on postoperative patient outcome. Moreover, metal ion levels will be measured in the blood stream preoperatively (as reference) and upon follow-up, based on previous observations that metal ion levels are increased in serum following TKA, without any relevant influence on outcome.

Aims

The aim of the present prospective study is to assess whether differences in tribological pairings - i.e. TiN-coating in comparison to CoCr-alloy using a frequently implanted total knee endoprosthesis (ACS® System, Implantcast GmbH, Buxtehude, Germany) - have an effect on postoperative range of motion (ROM) and patient satisfaction, reflected by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Forgotten Joint Score (FJS), Knee Society Score (KSS), Visual Analogue Scale (VAS). Moreover, metal ion levels will be tested in both groups to monitor their concentration in the blood stream, usually reflecting physiological abrasion.

Endpoints

The primary endpoint of the current study is the functional outcome of patients with TKA on a CoCrMo- basis in comparison to a TiN-coated implant. The secondary endpoint is the measurement of metal ion levels in the blood stream and their potential dynamics over time.

Methods

Two-hundred patients will be prospectively included in the study over a 4-year period, with 100 being randomly assigned to group A (TiN-coating) and 100 to group B (CoCr-alloy).

Random assignment will be carried out via an automatic randomisation system run by a local study nurse. Pre- and postoperatively, range of motion (ROM), visual analogue scale (VAS) score and specific questionnaires - i.e. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Forgotten Joint Score (FJS), Knee Society Score (KSS) - will be ascertained (Table 1) in order to allow comparison of potential differences between group A and B during follow-up. Furthermore, preoperatively, at 6 months, 12 months, 24 months and 60 months, metal ion levels (cobalt, chromium, molybdenum, titanium) in the blood stream will be measured in each patient (6ml tubes). Measurements of metal ion levels will be performed at an external institution.

The phase of active recruiting is planned for 4 years, with 50 patients being included per year on average. With the last patients anticipated to being included at the end of the 4th year, their follow-up will be finished 9 years after study initiation.

Randomisation and Blinding

All patients will be informed prior to potential study participation whether or not to they would like to participate, clarifying that refusal will not have any negative impact on further treatment. In case patients agree to participate, they will be randomly assigned to either group A or B.

Double-blinding will be made possible by not informing patients whether they had been allocated to group A or B and by not directly revealing information about the implant type used on medical records that will later be accessible to the study nurse and/or physicians during clinical examinations at follow- up. Therefore, it will be necessary to exclude those surgeons participating in the surgeries of the respective patients from examining them during follow-up, in order to maintain blinding. Prior to follow-up appointments, surgeons who had not participated in surgeries of the respective patients will thus be informed by the study nurse in order to perform clinical examination, radiological follow-up and questionnaires.

Expected Results

As patients receive the identical orthopaedic implant during an identical surgical procedure for comparable indications, it is expected that the differences in alloy (i.e. TiN vs. CoCr) will not have a measurable effect on postoperative patient outcome. Neither there is expected to be a difference in metal ion levels in the blood stream over time between groups.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis of index knee
* Varus angle < 15° of index knee

Exclusion Criteria:

* Previous native knee infection of index knee
* Previous distal femoral fracture of index knee
* Previous proximal tibial fracture of index knee
* Preceding osteotomy of index knee
* Known allergies against metals, drugs, organic substances
* Unicondylar prosthetic replacement of index knee
* Knee osteoarthritis of both joints with planned simultaneous TKA

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Change of Postoperative functional outcome - ROM with goniometer | Preoperatively, postoperative week 6, month 12, month 24, month 60.
  Range of motion (ROM), assessed with goniometer approved for medical issues
Change of Postoperative functional outcome - pain | Preoperatively, postoperative week 6, month 12, month 24, month 60.
  VAS score (Visual Analogue Scale; 0 = no pain, 10 = severe pain)
Change of Postoperative functional outcome - Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Preoperatively, postoperative week 6, month 12, month 24, month 60.
  Assessed by Western Ontario and McMaster Universities Arthritis Index (WOMAC). This index ranges from 0 to 100 points and is based on items pain, physical function and joint stiffness. Lower values indicating better outcomes, whilst higher values point towards worse outcome.
  Higher scores on the WOMAC indicate a worse outcome
Change of Postoperative functional outcome - FJS | Preoperatively, postoperative week 6, month 12, month 24, month 60.
  Forgotten Joint Score (FJS) with a scale ranging from 0 to 100, where a high value indicates a better outcome
Change of Postoperative functional outcome - Knee Society Score (KSS) | Preoperatively, postoperative week 6, month 12, month 24, month 60.
  Knee society score (KSS) is built up by two scores, i.e. "Functional Score" (3 items) and "Knee Score" (7 items), both ranging from 0 to 100 points. The lower the values, the worse the outcome.

SECONDARY OUTCOMES:
Change of Metal ion levels in blood stream | Preoperatively, month 6, month 12, month 24, month 60.
  Measurement of titanium, cobalt, chromium, molybdenum in blood stream at specific time-points.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics and Trauma, Medical University of Graz, Austria, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
It is not planned to share the IPD in full. However, results of the study are planned to be made public within a scientific work.

REFERENCES:
- [Background] Fabry C, Zietz C, Baumann A, Ehall R, Bader R. High wear resistance of femoral components coated with titanium nitride: a retrieval analysis. Knee Surg Sports Traumatol Arthrosc. 2018 Sep;26(9):2630-2639. doi: 10.1007/s00167-017-4578-7. Epub 2017 May 20. PMID 28528349
- [Background] Fennema P, Heyse TJ, Uyl-de Groot CA. Cost-effectiveness and clinical implications of advanced bearings in total knee arthroplasty: a long-term modeling analysis. Int J Technol Assess Health Care. 2014 Apr;30(2):218-25. doi: 10.1017/S0266462314000129. Epub 2014 Apr 28. PMID 24774225
- [Background] Gudnason A, Hailer NP, W-Dahl A, Sundberg M, Robertsson O. All-Polyethylene Versus Metal-Backed Tibial Components-An Analysis of 27,733 Cruciate-Retaining Total Knee Replacements from the Swedish Knee Arthroplasty Register. J Bone Joint Surg Am. 2014 Jun 18;96(12):994-999. doi: 10.2106/JBJS.M.00373. PMID 24951734
- [Background] Lapaj L, Wendland J, Markuszewski J, Mroz A, Wisniewski T. Retrieval analysis of titanium nitride (TiN) coated prosthetic femoral heads articulating with polyethylene. J Mech Behav Biomed Mater. 2015 Mar;55:127-139. doi: 10.1016/j.jmbbm.2015.10.012. Epub 2015 Oct 30. PMID 26584076
- [Background] Longo UG, Ciuffreda M, D'Andrea V, Mannering N, Locher J, Denaro V. All-polyethylene versus metal-backed tibial component in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3620-3636. doi: 10.1007/s00167-016-4168-0. Epub 2016 May 21. PMID 27209191
- [Background] Paxton EW, Inacio MC, Kurtz S, Love R, Cafri G, Namba RS. Is there a difference in total knee arthroplasty risk of revision in highly crosslinked versus conventional polyethylene? Clin Orthop Relat Res. 2015 Mar;473(3):999-1008. doi: 10.1007/s11999-014-4046-3. PMID 25567357
- [Background] Postler A, Beyer F, Lutzner C, Tille E, Lutzner J. Similar outcome during short-term follow-up after coated and uncoated total knee arthroplasty: a randomized controlled study. Knee Surg Sports Traumatol Arthrosc. 2018 Nov;26(11):3459-3467. doi: 10.1007/s00167-018-4928-0. Epub 2018 Apr 3. PMID 29616285